CLINICAL TRIAL: NCT01055184
Title: Assessment of the Effect of Age on the Immunological and Virological Response to a Live Attenuated Influenza Vaccine for the 2009 H1N1 Virus
Brief Title: Effects of Age on Response to the 2009 H1N1 Virus Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, John Treanor, M.D., University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URMC 09-009
Record Dates: First submitted 2010-01-05; First posted 2010-01-25 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: 2009 H1N1 Influenza Virus
Keywords: Influenza; H1N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2009 H1N1 Vaccine (Experimental): Participants will be stratified by age into two groups: those between 60 and 70 years old, and those older than 70 years of age. All participants will receive the 2009 H1N1 vaccine.
  Interventions: Biological: 2009 H1N1 Virus Vaccine

INTERVENTIONS:
Biological: 2009 H1N1 Virus Vaccine — Single 0.2 mL dose of live monovalent vaccine, delivered through nasal spray
  Other Names: Influenza A (H1N1) 2009 Monovalent Vaccine Live, Intranasal

SUMMARY:
Unlike most influenza viruses, the 2009 H1N1 virus has affected people between 5 and 40 years old more often than people 60 years old or older. It may be that older people have had greater exposure to previous strains of H1N1 influenza, and this previous exposure protects them from infection. This study will examine how older people respond to a version of the H1N1 virus vaccine that includes a live, noninfectious version of the virus.

DETAILED DESCRIPTION:
Unlike most influenza viruses, the 2009 H1N1 virus affects many individuals between 5 and 40 years old, but very few 60 years old or older. It is not completely understood why, but scientists believe it may be because older people may have been exposed to other H1N1 viruses in their lives. H1N1 viruses were common until 1957, when they were eclipsed by H2N2 viruses.

In order to test susceptibility to the 2009 H1N1 virus, this study will examine how often people older than 60 get infected by the 2009 H1N1 live attenuated influenza vaccine (LAIV). The LAIV is made from a live virus that has been weakened, so the ability of the immune system to combat this weakened form is likely to mimic its ability to combat the normal form. Additionally, this study will examine how LAIVs work in older people; inactivated virus vaccines are used more often than LAIVs in older people, so little is known of LAIV's effects on this population.

Participation in this study will last 6 months. Participants will be people older than 60, divided into equal groups of people between the ages of 60 and 70 and people older than 70. Both groups will receive one dose of LAIV for 2009 H1N1 vaccine.

There will be six study visits, occurring at baseline and 2, 5, 7, 28, and 180 days after vaccination. Nasal wicks and throat swabs will be taken on Days 2, 5, and 7; a nasal wick alone will be taken at baseline and on Day 28. Blood samples will be taken at baseline and on Days 7 and 28. Participants will undergo physical exams at each visit.

ELIGIBILITY:
Inclusion Criteria:

* No prior history of infection with novel H1N1 virus or immunization with novel H1N1 vaccine documented by a laboratory
* Female participants must not be capable of becoming pregnant or take steps to prevent pregnancy from 30 days before enrollment to 30 days after receiving the study vaccine
* In good health, as determined by medical history and targeted physical examination
* Able to understand and comply with the planned study procedures, including being available for all study visits

Exclusion Criteria:

* Pregnancy
* Previous history of vaccination against novel H1N1 virus or a laboratory documented history of previous novel H1N1 infection
* Immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs or use of anticancer chemotherapy or radiation therapy within the preceding 36 months
* Active neoplastic disease (excluding nonmelanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years.
* Long-term (greater than 2 weeks) use of oral or parenteral steroids or high-dose inhaled steroids (greater than 800 mcg/day of beclomethasone dipropionate or equivalent) within the 6 months prior to study enrollment (nasal and topical steroids are allowed)
* Received immunoglobulin or another blood product within the 3 months prior to enrollment in this study
* Received an inactivated vaccine within 2 weeks or a live vaccine within 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses.
* Has had an acute illness or an oral temperature greater than 99.9°F (37.7°C) within 3 days prior to enrollment or vaccination. Subjects who had an acute illness that was treated with symptoms resolved are eligible to enroll as long as treatment is completed and symptoms are resolved more than 3 days prior to enrollment.
* Currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication), has received an experimental agent within 1 month prior to enrollment in this study, expects to receive another experimental agent during participation in this study, or intends to donate blood during the study period
* History of alcohol or drug abuse in the 5 years prior to enrollment
* Has a known human immunodeficiency virus (HIV) or hepatitis B or C infection
* Has a previous history of Guillain-Barré syndrome
* Allergic to eggs or egg proteins, gentamicin, gelatin, or arginine or has experienced life-threatening reactions to previous influenza vaccination
* Has any other condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Vaccine Research Unit, Rochester, New York, United States

REFERENCES:
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216
- [Background] Cutler J, Schleihauf E, Hatchette TF, Billard B, Watson-Creed G, Davidson R, Li Y, Bastien N, Sarwal S; Nova Scotia Human Swine Influenza Investigation Team. Investigation of the first cases of human-to-human infection with the new swine-origin influenza A (H1N1) virus in Canada. CMAJ. 2009 Aug 4;181(3-4):159-63. doi: 10.1503/cmaj.090859. Epub 2009 Jul 20. PMID 19620268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were recruited from 3/24/2010 to 11/17/2010. Potential subjects were seen at the Vaccine research Unit clinic.
Pre-assignment Details: Only subjects who did not meet inclusion/exclusion criteria were excluded from participation.
Groups:
- 2009 H1N1 Vaccine: To ensure balance in the age distribution of the study, participants will be stratified by age into two groups: those between 60 and 70 years old, and those older than 70 years of age. All participants will receive the 2009 H1N1 vaccine.
Period: Overall Study
Arm/Group | 2009 H1N1 Vaccine
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2009 H1N1 Vaccine
Number analyzed (Participants) | 34
Age, Customized [Number; unit: participants]
  60-70 years | 20
  >70 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Shed Virus
Description: number of participants who shed virus above the limit of detection at any timepoint after vaccine. The limit of detection is 0.5 tissue culture infectious doses per mL of nasal wash.
Time Frame: day 0 to day 7 post vaccination
Measure: Number; unit: participants
Arm/Group | 2009 H1N1 Vaccine
Number analyzed (Participants) | 34
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from day 0 thru Dy 180
Arm/Group | 2009 H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2009 H1N1 Vaccine (N=34)
Aortic Stenosis (Cardiac disorders) | 1 (1) — Grade severe, Relationship - not associated, Subject recovered without sequelae
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2009 H1N1 Vaccine (N=34)
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 1, Relationship - associated, outcome resolved
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1, Relationship - not associated, Outcome resolved
Shingles (Infections and infestations) | 1 (1) — Grade 1, Relationship - not associated, Outcome resolved
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) — All events were Grade 1, Relationship not associated, Outcome resolved
Achy legs (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1, Relationship - associated, Outcome resolved
Ringing in ears (Ear and labyrinth disorders) | 1 (1) — Grade 1, Relationship - associated, Outcome recovered
Bone spurs left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 2, Relationship - not associated, Outcome recovered
Urinary Tract Infection (Infections and infestations) | 1 (1) — Grade 1, Relationship - not associated, Outcome recovered
Pinched nerve in neck (Nervous system disorders) | 1 (1) — Grade 2, Relationship - not associated, Outcome recovered
Lower back pain - left side (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1, Relationship - not associated, Outcome Recovered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No